CLINICAL TRIAL: NCT06461351
Title: A Long Term Follow-up Observational Study of Patients Treated With Inaticabtagene Autoleucel Injection
Brief Title: Long-term Observational Study of Patients Treated With Inaticabtagene Autoleucel Injection
Status: Recruiting | Type: Observational
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HY001401
Record Dates: First submitted 2024-06-06; First posted 2024-06-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: B-cell Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Inaticabtagene autoleucel Injection — Inaticabtagene autoleucel Injection
  Other Names: CNCT19

SUMMARY:
This clinical trial adopts an observational research method to conduct annual follow-up and monitoring of patients receiving treatment with Inaticabtagene Autoleucel Injection after its commercialization, in order to evaluate the delayed adverse events of Inaticabtagene Autoleucel Injection.

DETAILED DESCRIPTION:
Patients treated with Inaticabtagene Autoleucel Injection (including registered clinical trial patients with different indications of this product and commercialized patients after market launch), would be included in this program for a maximum of 15 years of long-term follow-up (LTFU), and an informed consent form must be signed again. The research period was 15 years after Inaticabtagene Autoleucel infusion. The patient was followed up once a year for 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to sign an informed consent form for long-term follow-up studies.
2. Registered clinical trial patients with different indications for this product who have received at least one infusion of Inaticabtagene Autoleucel Injection in the past, as well as post market commercialized patients.

Exclusion Criteria:

- None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registered clinical trial patients with different indications and post market commercialized patients who have received treatment with Inaticabtagene Autoleucel Injection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2039-05-30 (Estimated); Study Completion 2040-03-30 (Estimated)

PRIMARY OUTCOMES:
Replication-competent lentivirus，RCL | once a year from date of Inaticabtagene Autoleucel Injection treatment until date of death from any cause, assessed up to 15 years.
  Real time quantitative polymerase chain reaction was used for detection, QPCR method.

SECONDARY OUTCOMES:
Long-term Adverse Drug Reaction | once a year from date of Inaticabtagene Autoleucel Injection treatment until date of death from any cause, assessed up to 15 years.
  Individual adverse drug reactions related to Inaticabtagene Autoleucel Injection after marketing, mainly including secondary tumors, etc after marketing, mainly including secondary tumors, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Tianjin, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No